CLINICAL TRIAL: NCT05148104
Title: Intra-operative Evaluation of the Glenoid Implant Position With Structured Light
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Robin Richards, Orthopaedic Surgeon, Division of Orthopaedic Surgery, Sunnybrook Health Sciences Centre
Other Study IDs: Bullseye Glenoid
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving shoulder arthroplasty: Patients receiving shoulder arthroplasty that have an intact glenoid prior to the procedure. Ideally the glenoid surface should be visible and intact during imaging.

SUMMARY:
Positioning of the glenoid component is one of the most challenging steps in shoulder replacement surgery. Prosthesis longevity and functional outcomes are considered highly dependent on accurate positioning. Currently, there are no adequate means to verify the position of the glenoid component during surgery which is a significant impediment to accurate positioning. We propose a non-interventional study to validate a novel technology for verifying the position of the glenoid component during shoulder replacement surgery.

DETAILED DESCRIPTION:
Positioning of the glenoid component is one of the most challenging steps in shoulder replacement surgery. In this study, we are testing a new method of checking the glenoid component position using an optical light 3D scanner for both total and reverse total shoulder replacements. Currently, the position of the glenoid component is verified by the operating surgeon visually and there is no routine imaging to verify the position of the glenoid component during surgery.

Participants in this study will have a 3D optical image of their glenoid bone taken during the surgical procedure. Taking this image will require less than 3 minutes and the image will only include their surgical wound (no facial features or other identifying features will be taken in the images). Two to six weeks after the surgery, the study participants will have CT scan of their replaced shoulder. This will allow the researchers to measure the accuracy of the new imaging system.

It is anticipated that about 14 people will participate in this study at Sunnybrook. The length of this study for participants is 6 weeks. The entire study is expected to take about 1 year to complete and the results should be known 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* Scheduled to undergo total shoulder arthroplasty surgery.
* Scheduled pre-operative CT imaging of the shoulder and the surgical plan includes open exposure of the glenoid.

Exclusion Criteria:

* Previous shoulder surgery involving the glenoid.
* No clinically indicated pre-operative CT imaging.
* Pregnancy (current or planned).
* Current or planned participation in other research, or having a clinical condition that would result in cumulative annual radiation exposure exceeding the regulatory limit (30 mSv) from all sources.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be an eligible participant in this study, the patient must be about to undergo a total shoulder replacement.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Identify accuracy of the structured light computer vision system | Surgical timepoint
  The primary study outcome will be the accuracy of the structured light computer vision system. The outcome is a single measure quantified by the difference in predicted and actual position of the glenoid implant. The measure of the difference is a combination of version error (degrees), inclination error (degrees), and offset error (mm).

SECONDARY OUTCOMES:
Operative delay for imaging (seconds) | Surgical timepoint
  seconds
Computer vision system image processing time (seconds) | Surgical timepoint
  seconds
Intra-operative complications | Surgical timepoint
  from chart review
Early post-operative complications (evaluated at 3 months follow-up from chart review) | 3 months after surgery
  from chart review

CONTACTS AND LOCATIONS:
Overall Officials: Robin R Richards, MD, Principal Investigator — Appointed Orthopaedic Surgeon
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No